CLINICAL TRIAL: NCT03693976
Title: Non-interventional Study in Patients With Acute Rhinosinusitis to Study Efficacy and Tolerability of Ectoin Rhinosinusitis Nasal Spray, a Xylometazoline-containing Nasal Spray or a Combination of Both.
Brief Title: Non-interventional Study With Ectoin Containing and/or Decongesting Nasal Spray in Patients With Rhinosinusitis
Status: Completed | Type: Observational
Sponsor: Bitop AG (Industry)
Responsible Party: Sponsor
Other Study IDs: btph-010-2018-SNS01
Record Dates: First submitted 2018-10-01; First posted 2018-10-03 (Actual); Last update posted 2019-07-10 (Actual); Status verified 2018-11

CONDITIONS: Acute Rhinosinusitis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Ectoin Rhinosinusitis Nasal Spray: application of 1-2 sprays of SNS01 into each nostril several times a day
  Interventions: Device: Ectoin Rhinosinusitis Nasal Spray
- Xylometazoline nasal spray: 1 spray per nostril as often as required but not exceeding 3 sprays per nostril per day
  Interventions: Drug: Xylometazoline Nasal Spray
- Xylometazoline + Ectoin Nasal Spray: Xylometazoline: 1 spray per nostril as often as required but not exceeding 3 sprays per nostril per day, Ectoin Nasal Spray (SNS01): 1-2 sprays per nostril several times a day
  Interventions: Drug: Xylometazoline Nasal Spray; Device: Ectoin Rhinosinusitis Nasal Spray

INTERVENTIONS:
Drug: Xylometazoline Nasal Spray — Application of Xylometazoline Nasal Spray in accordance with the instructions for use
  Other Names: NasenSpray-ratiopharm Erwachsene (adults)
  Groups: Xylometazoline + Ectoin Nasal Spray; Xylometazoline nasal spray
Device: Ectoin Rhinosinusitis Nasal Spray — Application of Ectoin Nasal Spray (SNS01) in accordance with the instructions for use
  Other Names: SNS01
  Groups: Ectoin Rhinosinusitis Nasal Spray; Xylometazoline + Ectoin Nasal Spray

SUMMARY:
The goal of this non-interventional study is to investigate the efficacy and tolerability of an Ectoin containing Rhinosinusitis Nasal Spray (SNS01). Within the study, SNS01 will be used either alone as monotherapy or as concomitant therapy in addition to the use of a Xylometazoline-containing decongestant nasal spray. A control group will use a Xylometazoline-containing decongestant nasal spray as monotherapy.

It will be investigated if the dose of the used decongestant nasal spray might be reduced, the development of the disease might be positively influenced and/or the potentially occurring side effects (e.g. dryness of the nasal mucosa, sneezing) might be alleviated by using the Ectoin containing Rhinosinusitis Nasal Spray as concomitant therapy.

DETAILED DESCRIPTION:
The current non-interventional study aims to investigate the efficacy and tolerability of Ectoin containing Rhinosinusitis Nasal Spray (SNS01) in patients with acute rhinosinusitis. Patients can chose one of three treatment options: a) Ectoin containing Rhinosinusitis Nasal Spray (SNS01), b) decongestant Xylometazoline-containing nasal spray or c) Ectoin containing Rhinosinusitis Nasal Spray (SNS01) and a decongestant Xylometazoline-containing nasal spray.

Efficacy will be studied by documentation of the following symptoms:

* oedema, redness (assessed by rhinoscopy)
* nasal obstruction, nasal secretion, headache/face pain, loss of sense of smell/taste
* sore throat, cough

In parallel, participating patients will document their symptoms and the their quality of life over the entire study duration in patient diaries.

Patients of both genders aged 6 years and above can take part in the study if diagnosed with acute viral rhinosinusitis. The assignment of a patient to a particular treatment is not decided in advance but falls within current practice, and is clearly separated from the decision to include the patient into the study.

Study therapy will be applied in accordance with the respective instructions for use.

Study duration is 7-14 days, depending on the improvement of symptoms. At the end of the study, both the investigators and the patients are asked to judge the efficacy and tolerability of the treatments.

ELIGIBILITY:
Inclusion Criteria:

* patients with acute viral rhinosinusitis
* presence of common cold symptoms

Exclusion Criteria:

* contraindications in accordance with instructions for use
* acute bacterial rhinosinusitis
* chronic rhinosinusitis

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients aged above 6 years diagnosed with acute viral rhinosinusitis
Sampling Method: Non-Probability Sample
Enrollment: 168 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2019-04-15 (Actual); Study Completion 2019-04-15 (Actual)

PRIMARY OUTCOMES:
Physicians' assessment of change of intensity of rhinosinusitis symptoms | day 0 and day 7 and (if necessary, depending on study duration) and on day 14
  Both on day 0 and on day 7 (and, if necessary, depending on study duration, on day 14), the physicians will assess rhinosinusitis symptoms oedema, redness of the nose, nasal obstruction, nasal secretion, facial pain/headache, smell/taste dysfunction and the concomitant symptoms dryness of the nasal mucosa and sore throat. Assessment will be carried out based on a 5-point scale (0=none to 4=very strong). Change of symptoms will be assessed comparing symptom scores on day 7 (or day 14, if applicable) to day 0. The investigators will use rhinoscopy, physical examination and interview of the patients for the assessments.

SECONDARY OUTCOMES:
Physicians' assessment of general well-being of patients | day 0 and day 7 and day 14 (if necessary, depending on study duration)
  The investigators will assess the well-being of patients using a 4-point scale (good condition to strong illness).
Patients' assessment of intensity of symptoms and their influence on quality of life | 7 to 14 days (depending on study duration)
  Patients will document their rhinosinusitis symptoms and their influence on quality of life (22 parameters in accordance with the "sino-nasal outcome test-22 questionnaire") and the additional symptom "dry nose". They will document their judgement daily in a patient diary using a 6-point scale (0=no problem to 5=as bad as possible).
Investigators' and patients' assessment of efficacy of treatments | once on day 7 or day 14 (depending on study duration)
  At the end of the study, both investigators and patients will judge the overall efficacy of the treatment based on a 6-point scale (1=very good to 6=unsatisfactory).
Assessment of the tolerability of treatments | once on day 7 or once on day 14 of treatment (depending on study duration)
  Both investigators and patients will judge the tolerability of the treatments at the end of the study. Both investigators and patients will judge the tolerability based on a 6 point scale (1=very good to 6 = unsatisfactory).
Incidence of adverse events/serious adverse events | 7 to 14 days (depending on study duration)
  All occurring adverse events/serious adverse events will be documented during the entire study period.

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Bilstein, Dr., Study Director — CSO
Locations (1):
- bitop AG, Dortmund, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Werkhauser N, Bilstein A, Mahlstedt K, Sonnemann U. Observational study investigating Ectoin(R) Rhinitis Nasal Spray as natural treatment option of acute rhinosinusitis compared to treatment with Xylometazoline. Eur Arch Otorhinolaryngol. 2022 Mar;279(3):1371-1381. doi: 10.1007/s00405-021-06916-0. Epub 2021 Jun 4. PMID 34089097